CLINICAL TRIAL: NCT07236957
Title: Corrected Weight to the 10th Percentile vs. Actual Birth Weight for the Calculation of Nutritional Needs of Small for Gestational Age Neonates Fed on Parenteral Nutrition: a Randomized-controlled Trial
Brief Title: Estimation of Nutritional Needs of Preterm Neonates Fed on Parenteral Nutrition and Effects on Body Weight Gain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Panos Papandreou (Other)
Collaborators: University of Peloponnese (Other)
Responsible Party: Sponsor-Investigator, Panos Papandreou, Head Pharmacologist, Iaso Maternity Hospital, Athens, Greece
Organization: Iaso Maternity Hospital, Athens, Greece (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 21-11-18AB
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Preterm Infant Development; Preterm Infant Feeding Outcomes
Keywords: preterm neonates; parenteral nutrition; clinical decision support system; weight gain
MeSH Terms: conditions — Hyperphagia; Weight Gain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A total of 100 preterm and small for gestational age neonates were randomly assigned to either the Control group (n = 50) or the Intervention group (n = 50). Both groups received parenteral nutrition (PN) supported by a specialized clinical decision support system. In the Control group, the PN regimen was based on the actual birth weight, whereas in the Intervention group, calculations were based on the corrected weight corresponding to the 10th percentile of the growth curve.
Who Masked: Care Provider
Masking Description: The care providers who administered the parenteral (PN) solutions to the neonates were blinded to the identity of the PN solution.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutrient estimation based on the actual weight (Control group) (Sham Comparator): In the Control group, the clinical decision support system was used to determine parenteral nutriton requirements.
  Interventions: Dietary Supplement: Control group
- Nutrient estimations based on the corrected weight (Intervention group) (Active Comparator): In the Intervention group, the clinical decision support system was used to determine parenteral nutrition requirements.
  Interventions: Dietary Supplement: Intervention Group

INTERVENTIONS:
Dietary Supplement: Intervention Group — In the Intervention group, the macronutrient composition in the parenteral nutrition solutions was calculated based on the corrected weight corresponding to the 10th percentile of the growth curve.
  Arms: Nutrient estimations based on the corrected weight (Intervention group)
Dietary Supplement: Control group — In the Control group, the parenteral nutrition regimen was estimiated based on the actual birth weight.
  Arms: Nutrient estimation based on the actual weight (Control group)

SUMMARY:
This randomized controlled trial included 100 preterm and small for gestational age neonates. The study aimed to determine the optimal approach for estimating nutritional needs in parenteral nutrition (PN) with the assistance of a specialized clinical decision support system (CDSS). More specifically, nutrient estimations based on the neonates' actual birth weight were compared to those calculated using the weight corresponding to the 10th percentile of the growth curve. The effect on growth outcomes over the PN course was investigated.

DETAILED DESCRIPTION:
Background: Parenteral nutrition (PN) plays a crucial role in providing nutritional support to premature and small for gestational age neonates.

Aim: In this randomized controlled study, we evaluated PN administration in preterm and small for gestational age neonates using the corrected weight estimated at the 10th percentile of the growth curve, as guided by a clinical decision support system (CDSS).

Methods: A total of 100 preterm neonates were randomly assigned to either the Control group (n = 50) or the Intervention group (n = 50). Both groups received PN support using a specialized CDSS. In the Control group, the CDSS calculated the PN regimen based on the actual birth weight, whereas in the Intervention group, calculations were based on the corrected weight corresponding to the 10th percentile. Growth indicators (i.e., body weight, length, and head circumference) were measured at baseline and at the time of exclusive enteral feeding initiation. Blood samples were obtained at the last day of PN, after PN was ceased for 4 h and before oral feeding initiation. Electrolytes (sodium, potassium, calcium) and albumin concentrations, as well as red blood cells, white blood cells, haemoglobin and haematocrit were measured at the last day of PN.

ELIGIBILITY:
Inclusion Criteria:

* preterm neonates hospitalized in NICU and meeting the criteria for small for gestational age infants, i.e., neonates with birth weight under the 10th percentile,
* preterm neonates receiving exclusive parenteral nutrition, and
* parents' written consent for study participation.

Exclusion Criteria:

* term birth newborns or newborns not fullfilling the criteria of small for gestational age infants,
* newborns with primary liver/bile duct disease,
* newborns receiving enteral nutrition, and/or
* neonates whose parents did not give a written consent to participate in the study

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Body weight change | From birth day (day 1) till the last day of parenteral nutrition support (study endpoint). Each neonate had different PN duration according to their clinical status (average 12 days).
  The primary outcome is to detect a statistical significant difference in body weight increase between the control and the intrevention group at the last day of parenteral nutrition support (study endpoint).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, IASO Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available on request from the corresponding author. The data are not publicly available due to their containing information that could compromise the privacy of the research participants.

REFERENCES:
- [Background] Fenton TR, Kim JH. A systematic review and meta-analysis to revise the Fenton growth chart for preterm infants. BMC Pediatr. 2013 Apr 20;13:59. doi: 10.1186/1471-2431-13-59. PMID 23601190
- [Derived] Papandreou P, Foscolou A, Bampoukli E, Gioxari A. Parenteral nutrition using corrected weight to the 10th percentile improves weight gain in preterm neonates: a randomized controlled trial. Clin Nutr ESPEN. 2026 Feb 5:102960. doi: 10.1016/j.clnesp.2026.102960. Online ahead of print. PMID 41654298